CLINICAL TRIAL: NCT04254588
Title: Can Telemedicine Examinations of the Abdomen Safely Determine the Need for Abdominal Imaging?
Brief Title: Telemedicine Abdominal Exams & Imaging
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Crico (Other)
Responsible Party: Principal Investigator, Emily Marie Hayden, Attending Physician and Director of Telemedicine, Department of Emergency Medicine, Massachusetts General Hospital
Other Study IDs: 2018P002608
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Abdominal Pain
Keywords: Emergency Department, Telemedicine, Telehealth
MeSH Terms: conditions — Abdominal Pain; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase I: Adult patients with abdominal pain: Adult patients with abdominal pain presenting to the MGH ED between February and March 2020.
  Interventions: Other: Abdominal examination
- Phase II: Adult patients with abdominal pain: Adult patients with abdominal pain presenting to the MGH ED between July and December 2021.
  Interventions: Other: Abdominal examination

INTERVENTIONS:
Other: Abdominal examination — Examination by in-person physician vs. remote physician.

SUMMARY:
A study of patients with abdominal pain being seen by physicians at an academic emergency department and by physicians who are based remotely (telehealth).

Hypothesis: When a patient with abdominal pain is examined by a physician at the hospital versus a physician who is remote (i.e. not at the hospital), they will agree most of the time for the need of abdominal imaging for the patient within 12 hours of their examination.

DETAILED DESCRIPTION:
This will be a prospective, observational, blinded diagnostic concordance study of patients being seen for abdominal pain at an academic emergency department (ED) at Massachusetts General Hospital (MGH).

The study will consist of two phases. Both phases will have an on-call telemedicine physician who will assess the patient and answer the question about need for imaging.

The first phase mitigates technical issues with the telemedicine technology by using the high-resolution MGH TeleHealth Stroke Cart. This will allow telemedicine hardware that has been vetted in the high-acuity and high-reliability Acute Stroke Service and will minimize the impact of potential technical problems with iPads and wireless connectivity.

The second phase will substitute the Stroke Cart with an iPad to mimic the devices that the patients will likely be using from home in a direct-to-patient telehealth program.

Initially, we expected to enroll up to 72 subjects in 2 phases. Each phase would have needed 30 patients for significant results, and another 6 patients are estimated for patients that may become ineligible during the study visit (e.g., potential for contamination if the subject mentions the abdominal imaging plans of the in-person provider during the telemedicine examination). Phase 1 provided more information and changed our assumptions for Phase 2 sample size. We increased Phase 2 enrollment target to 60 subjects; we need 53 patients for significant results and will add 7 patients should they become ineligible during the study. Therefore, a total of 90 subjects in Phase 1 and 2 will be enrolled.

After consent, the research staff member will page the on-call study telemedicine physician and bring the stroke cart (iPad in the second phase) into the examination room. The on-call physician will connect to the secure video application and will interview and examine the patient. The telemedicine physician will not tell the patient their thoughts on what is the cause of their pain, nor tell the patient the next steps in their care. The physician will thank the patient for their time and log off of the video call. The telemedicine provider will not place orders for the patient's emergency department visit, nor will they document in the patient's chart in the electronic medical record. The telehealth provider will only perform a telehealth-based examination and answer the study questions asked by the research staff member; all responses will be recorded on the electronic data capture (EDC) system. The research staff member will notify the in-person team that the telehealth examination is complete.

The in-person examination will follow the current standard of practice with the emergency physician scheduled for that shift. The research staff member will ask the same questions to the in-person provider after their examination and record the data on the EDC.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting to the MGH Emergency Department with abdominal pain
* English-speaking

Exclusion Criteria:

* Known to be pregnant
* Patients with altered mental status
* Patients who are critically ill or unstable

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: English-speaking patients >19 years of age, presenting to the MGH Emergency Department with abdominal pain will be eligible for the study. Women who are known to be pregnant will be excluded from the study. Patients will be excluded from the study if they have altered mental status or who are critically ill or unstable. Altered mental status patients will be excluded because they would not be able to consistently participate in a patient-assisted physical examination by following the provider's verbal directions. Critical illness or patients who are unstable will be excluded from the study if they are triaged to the critical care area (Acute) of the MGH Emergency Department.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Requirement of imaging after abdominal examination | 12 hours
  Questionnaire agreement (yes no) between the in-person and telehealth physicians for the requirement of imaging after abdominal examination.

CONTACTS AND LOCATIONS:
Overall Officials: Emily M Hayden, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to make individual participant data (IPD) available to other researchers.